CLINICAL TRIAL: NCT02834767
Title: Genioglossus Muscle Training for Snoring and Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: IRB201600916
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Snoring; Sleep Apnea, Obstructive
MeSH Terms: conditions — Snoring; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Group 1 Primary Snoring Treatment (Experimental): Intervention: Eight weeks of supervised use of the genioglossus muscle strength trainer. Training will occur 5 days per week for 8 weeks. Each daily training regimen to consist of 5 sets of 5 repetitions (25 repetitions total daily) of tongue contractions using the device.
  Interventions: Device: Genioglossis Strength Trainer
- Group 2 Primary Snoring Placebo (Placebo Comparator): Intervention: Eight weeks of supervised use of the placebo genioglossus muscle strength trainer. Training will occur 5 days per week for 8 weeks. Each daily training regimen to consist of 5 sets of 5 repetitions (25 repetitions total daily) of tongue contractions using the device.
  Interventions: Device: Placebo Genioglossis Strength Trainer
- Group 3 Primary OSA Treatment (Experimental): Intervention: Eight weeks of supervised use of the genioglossus muscle strength trainer. Training will occur 5 days per week for 8 weeks. Each daily training regimen to consist of 5 sets of 5 repetitions (25 repetitions total daily) of tongue contractions using the device.
  Interventions: Device: Genioglossis Strength Trainer
- Group 4 Primary OSA Placebo (Placebo Comparator): Intervention: Eight weeks of supervised use of the placebo genioglossus muscle strength trainer. Training will occur 5 days per week for 8 weeks. Each daily training regimen to consist of 5 sets of 5 repetitions (25 repetitions total daily) of tongue contractions using the device.
  Interventions: Device: Placebo Genioglossis Strength Trainer

INTERVENTIONS:
Device: Genioglossis Strength Trainer — The genioglossis strength trainer is a handheld device, manufactured in house, consisting of an outer tube, inner piston, and pressure loaded spring. The device can be set to a specific pressure resistance ranging from 10 to 40 Newtons. Users press against the inner piston with their tongues until the piston moves approximately 1/2 centimeter (and the inner pressure loaded spring depresses approximately 1/2 centimeter).
  Other Names: Tongue Strength Trainer
  Arms: Group 1 Primary Snoring Treatment; Group 3 Primary OSA Treatment
Device: Placebo Genioglossis Strength Trainer — The placebo genioglossis strength trainer is a handheld device, manufactured in house, consisting of an outer tube, inner piston, and pressure loaded spring. Whereas the pressure loaded spring in the active trainer can be set to a wide range of pressures, the placebo trainer has a maximum resistance of 5 Newtons. The device is set to a specific pressure resistance of 5 Newtons at all times. Users press against the inner piston with their tongues until the piston moves approximately 1/2 centimeter (and the inner pressure loaded spring depresses approximately 1/2 centimeter).
  Other Names: Placebo Tongue Strength Trainer
  Arms: Group 2 Primary Snoring Placebo; Group 4 Primary OSA Placebo

SUMMARY:
Obstructive sleep apnea (OSA) carries serious health consequences for patients. Evidence exists that some behavioral (e.g. exercise based) therapies may assist in lessening the severity of this disorder. The proposed investigation will examine the effects of eight weeks of genioglossus muscle strength training on measures of snoring and OSA severity as well as genioglossus protrusive muscle strength.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common disorder characterized by intermittent narrowing or closure of the upper airway during sleep. Loss of muscle tone with sleep onset and decreases in ventilatory drive following the loss of the wakefulness stimuli to breathe combine to result in upper airway closure in patients with structurally susceptible upper airways. The genioglossus (GG, tongue) muscle plays an important role in maintaining upper airway patency. The GG is responsible for tongue protrusion and stiffens the tongue and prevents posterior tongue displacement and upper airway closure. The GG is a phasic respiratory muscle. One can demonstrate inspiratory bursts in GG EMG activity slightly preceding the onset of inspiratory activity of respiratory pump muscles. The inspiratory bursts of GG activity also increase in response to negative pressure in the upper airway to help maintain upper airway patency. In some OSA patients this response is blunted. While one study did not find a difference in protrusion muscle strength between a group of OSA patients (apnea hypopnea index, AHI = 20/hour) and normal controls (Mortimore et al) there was wide variability in muscle strength at similar AHI values. Another study (Oh et al) did find a correlation between tongue protrusion strength and the apnea index (lower strength, higher apnea index). It is hypothesized that strength training of the GG will reduce snoring and sleep apneas by augmenting the resting GG tone and enhancing the ability of the muscle to respond to negative upper airway pressure. Training of upper airway muscles including the tongue is often used in rehabilitation of patients with prior cerebrovascular accidents or damage due to surgical resection for cancer. Typically, the patient presses the tongue against the back of the upper teeth (direction both upward and forward). However, it is believed that tongue protrusion is best trained by active forward protrusion of the tongue between the teeth under load. To facilitate GGs training participants will push a spring loaded piston forward with the tongue. The piston fits inside an outer chamber. The piston can also be connected to a force measuring device to estimate protrusive tongue force.

Two groups of participants will be examined: Group 1: primary snoring and Group 2: mild to moderate OSA patients (apnea-hypopnea index < 30/hour) who are not severely obese (BMI < 40 Kg/M2) and do not have significant structural abnormalities of the upper airway or muscle dysfunction. This preliminary investigation consists of a randomized controlled trial (training versus sham training) with two months of daily training (5 out of 7 days each week). A home sleep study (including EEG) will be performed before and following the training. The change in the apnea-hypopnea index adjusted for sleep stage and body position will be compared. Use of home sleep studies will dramatically reduce the cost of the study. A sleep technologist will educate subjects on performance of training maneuvers and meet with them weekly to observe the subject's technique and measure tongue strength. A training log will be kept by the subjects using training schedule sheets and training will be directly monitored at least 2 times weekly through with a study clinician (electronically via facetime, skype or by direct observation).

ELIGIBILITY:
Inclusion Criteria:

* Snoring + AHI < 5/hr (primary snoring group)
* AHI ≥ 5/hour and less than 30/hour (OSA group)
* Ability to understand and perform training.
* Ability to return to the UF Health Sleep Center 1X per week for the (8 week) duration of the study.

Exclusion Criteria:

* Pregnancy
* Prior Upper airway surgery (nasal surgery is allowed)
* Severe nasal obstruction
* BMI > 40 kg/M2
* Use of CPAP > 12 cm H2O *
* Use of potent narcotics
* History of arrhythmia (other than PACs and PVCs)
* Coronary artery disease or congestive heart failure (patients with controlled hypertension will be included),
* Moderate to severe lung disease
* History of pneumothorax.
* severe daytime sleepiness (falling asleep while driving or Epworth Sleepiness Scale > 14),
* History of chronic short sleep duration (< 5 hours).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-05-04 (Actual); Study Completion 2019-05-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tongue Pressure Force (MTPF) | Pre to post treatment (approximately 10 weeks)
  Maximum pressure generated (in Newtons) during tongue protrusion

SECONDARY OUTCOMES:
Snoring Severity | Pre to post treatment (approximately 10 weeks)
  Snoring sensor recording snoring frequency and amplitude during sleep
Apnea-Hypopnea Index | Pre to post treatment (approximately 10 weeks)
  Episodes of apnea and/or hypopnea scored during the course of sleep study

CONTACTS AND LOCATIONS:
Overall Officials: Richard Berry, M.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida Sleep Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No